CLINICAL TRIAL: NCT00965536
Title: A Local Non Interventional Retrospective Register Study of the Current Clinical Treatment Practices and the Number of Hospitalization Days With Seroquel or Seroquel Prolong.
Brief Title: Nis Register Study Comparing Seroquel and Seroquel Prolong
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NFI-SER-2009/1
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Comparing Hospitalisation Time With Seroquel and Seroquel Prolong
Keywords: Schizophrenia; Bipolar Disorder; Manic Disorder; Register study; Quetiapine; Quetiapine Prolong; Seroquel; Seroquel Prolong; Seroquel XR; In-patient
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Seroquel
- 2: Seroquel Prolong

SUMMARY:
The general aim of this non interventional study is to clarify what are the current clinical treatment practices of Quetiapine Immediate Release and Quetiapine Extended Release. The primary objectives of the study are:1.To collect information on the used Quetiapine Immediate Release or Quetiapine Extended Release medication 2.To collect information on duration and number of hospitalisation days 3.Change of GAF points

ELIGIBILITY:
Inclusion Criteria:

* Medication: Seroquel or Seroquel Prolong
* Diagnosis: F20-F29 or F30-F31 (ICD-10)
* In-patient

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: South Karelia Central Hospital in-patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hospitalisation time | 2008-2010
Treatment practice | 2008-2010

SECONDARY OUTCOMES:
Primary diagnosis | 2008-2010
Medication at the end of hospitalisation | 2008-2010
GAF rating points | 2008-2010

CONTACTS AND LOCATIONS:
Overall Officials: Yrjö Ovaskainen, Study Director — Medical Affairs Manager, MD, psychiatrist; Kari Hänninen, Principal Investigator — MD, psychiatrist
Locations (1):
- Research Site, Lappeenranta, Finland